CLINICAL TRIAL: NCT01897870
Title: The Effect of a Home-based Community Pharmacist-led Medication Management Program (HomeCoMe-program) Complementary to an In-hospital Medication Reconciliation Program on Drug-related Problems Post-discharge: A Prospective Cohort Study.
Brief Title: The Effect of a Pharmacist Home Visit on Drug-related Problems Post-discharge.
Acronym: HomeCoMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H.T. Ensing, PharmD, MSc (Other)
Collaborators: Zorggroep Almere (Other); Flevoziekenhuis (Other)
Responsible Party: Sponsor-Investigator, H.T. Ensing, PharmD, MSc, PharmD, MSc, Zorggroep Almere
Organization: Zorggroep Almere (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ZGA-1
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Adverse Drug Event; Readmission; Patient Compliance
Keywords: continuity of care; medicines management; home visit; drug-related problems
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HomeCoMe-program group (Experimental): the arm receiving the pharmacist home visit
  Interventions: Behavioral: HomeCoMe-program

INTERVENTIONS:
Behavioral: HomeCoMe-program — A home visit by patients own community pharmacist within seven days after hospital discharge. The community pharmacist will perform a semi-structured interview on (1) use of the prescribed medication, (2) ADEs, (3) adherence issues, by (A) assessing patient's needs and concerns around his pharmacotherapy, (B) identifying and solving obstacles for medicines intake, (C) checking on the need for a compliance aid, (D) collecting spare medication and finally (4) knowledge on medication use, when to take which medicine and why, and medication changes made during the hospitalisation.

SUMMARY:
the purpose of this study is to determine the the effect of a home-based medication management program on drug-related problems post-discharge.

DETAILED DESCRIPTION:
Inaccuracy of medication histories and lack of knowledge on actual medication use results in confusion about medication regimens and medication mismanagement before- during - and after hospital admission. This phenomenon accounts for many readmissions, longer duration of admission and preventable and serious Adverse Drug Events (ADEs) as a result of Drug Related Problems (DRPs). Several studies show that discharge medication reconciliation (MR) and counseling by a pharmacy employee reduces the amount of discrepancies in the discharge prescription lists. Still, no unequivocal effect of MR on the occurrence of DRPs after discharge has been shown. This is due to a shift in underlying potential harmful discrepancies from mainly patient based (unintended nonadherence) to mainly system based (eg dispensing errors) and might be explained by (1) suboptimal transfer of information (2) an overload of information during a stressful situation and (3) difficulty to implement changes in medication at home. Therefore the reduction of DRPs, improvement of patients' medication knowledge and initial adherence can probably most effectively be addressed in a multifaceted integrated transmural intervention. Repetition of important information is the key to success. Moreover, the first weeks following hospital discharge are most crucial in preventing drug-related problems as patients could slip back in old medication schemes, or new problems may arise, such as emerging ADEs due to medication changes made during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* patient uses more than three prescribed systemic drugs intended for chronic use at admission and discharge
* patient has an expected length of stay of 48 hours or longer

Exclusion Criteria:

* Patients admitted for scheduled chemotherapy
* Patients admitted for radiation therapy
* Patients admitted for transplantation
* Patients transferred from another hospital
* Patients transferred from another non-eligible ward within the same hospital
* No informed consent signed
* A live expectancy less than 6 months
* Inability to be counselled (e.g. cognitive dysfunction, language constraints who cannot be solved with an interpreter)
* Discharge to a nursing home (presuming dependence on medication administration)
* If patients' community pharmacy is not participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Identifying and solving adverse drug events (ADEs) and other drug-related problems (DRPs) post-discharge | within 7 days post-discharge
  The total number of assessed and solved ADEs post-discharge will be measured. Assessing and solving ADEs takes place during the pharmacist home visit.
  Using START-STOPP criteria on patients medication records, ADEs will also be compared between the intervention and usual care group.

SECONDARY OUTCOMES:
Improvement of adherence to medication at hospital discharge | up to 6 months after discharge
  The "medication possession ratio" will be calculated retrospectively from pharmacy dispensing data after 6 months to investigate patient's adherence and compared between the intervention and control group.
Patient assessment of medication knowledge at time of home visit | within 7 days after discharge
  At time of the home visit patients are asked about their knowledge (e.g. indication, dose regime, etc) regarding the medication they are taking. Knowledge is scored and lack of knowledge is solved by teaching the patient.
Types of interventions made at the pharmacist home visit | within 7 days after discharge
  The types of intervention the pharmacist works on during the 7 day follow-up home visit are assessed.
Patient satisfaction with the pharmacist home visit | Immediately after receiving the home visit
  The satisfaction survey consists of 13 interview questions, where the subject subjectively scores each question on a four-point scale, developed specifically for this study.
Assessment of patient reported health rating | at 14 days after discharge
  Patient are asked by telephone to report their health on a scale from 1 (worst imaginable health) to 10 (best imaginable health). Number are compared between the intervention and control group.
General practitioners satisfaction with the pharmacist home visit | Immediately after the home visit is executed
  The satisfaction survey consists of 13 interview questions, where the subject subjectively scores each question on a four-point scale, developed specifically for this study.
Assessment of patient reported health rating | at 42 days after discharge
  Patient are asked by telephone to report their health on a scale from 1 (worst imaginable health) to 10 (best imaginable health). Number are compared between the intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel L Bouvy, Prof, PharmD, PhD, Principal Investigator — UIPS
Locations (1):
- Zorgapotheken Flevoland, Almere Stad, Flevoland, Netherlands

REFERENCES:
- [Background] Schnipper JL, Kirwin JL, Cotugno MC, Wahlstrom SA, Brown BA, Tarvin E, Kachalia A, Horng M, Roy CL, McKean SC, Bates DW. Role of pharmacist counseling in preventing adverse drug events after hospitalization. Arch Intern Med. 2006 Mar 13;166(5):565-71. doi: 10.1001/archinte.166.5.565. PMID 16534045
- [Background] Al-Rashed SA, Wright DJ, Roebuck N, Sunter W, Chrystyn H. The value of inpatient pharmaceutical counselling to elderly patients prior to discharge. Br J Clin Pharmacol. 2002 Dec;54(6):657-64. doi: 10.1046/j.1365-2125.2002.01707.x. PMID 12492615
- [Background] Kwint HF, Faber A, Gussekloo J, Bouvy ML. The contribution of patient interviews to the identification of drug-related problems in home medication review. J Clin Pharm Ther. 2012 Dec;37(6):674-80. doi: 10.1111/j.1365-2710.2012.01370.x. Epub 2012 Aug 3. PMID 22861493